CLINICAL TRIAL: NCT00305305
Title: Disorders of Cerebral Development: A Phenotypic and Genetic Analysis
Brief Title: Brain Development Research Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Washington (Other); California Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: UCSF-PCRC #2206
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Brain Disorders; Aicardi Syndrome
Keywords: Agenesis Corpus Callosum; Polymicrogyria; Dandy-Walker; Brain Malformation; Autism; Epilepsy; Mental Retardation; MRI; Agenesis of the Corpus Callosum (complete or partial); Confirmed by a brain MRI.; Aicardi Syndrome.
MeSH Terms: conditions — Brain Diseases; Aicardi Syndrome; Agenesis of Corpus Callosum; Polymicrogyria; Autistic Disorder; Epilepsy; Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Dr. Elliott Sherr and his collaborators at University of California, San Francisco (UCSF) are studying the genetic causes of disorders of cognition and epilepsy, in particular disorders of brain development that affect the corpus callosum, such as Aicardi syndrome, as well as two additional brain malformations, polymicrogyria and Dandy-Walker malformation. The goal of the investigators' research is to use a better understanding of the underlying genetic causes as a foundation to develop better treatments for these groups of patients.

DETAILED DESCRIPTION:
We are studying both the genetics and clinical features of these disorders. We hope to understand the problems faced by individuals with these disorders as well as their causes. In the future, we hope to develop therapies that are geared specifically for individuals based on the underlying biology. To participate in the study, you will be asked to provide a copy of the magnetic resonance imaging (MRI) documenting Agenesis Corpus Callosum (ACC), Polymicrogyria (PMG), or Dandy-Walker malformation (DWM), clinical information, and saliva or blood samples from the affected individual and from the parents. Please see contact information and our webpage below.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of agenesis or dysgenesis of the corpus callosum, polymicrogyria, or Dandy-Walker malformation
* Should be confirmed by an MRI (Magnetic Resonance Imaging) of the brain

Exclusion Criteria:

* Fully formed but hypoplastic corpus callosum

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with agenesis or dysgenesis of the corpus callosum, polymicrogyria, or cerebellar hypoplasia.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2003-08; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott H Sherr, MD, PhD, Principal Investigator — University of California, San Francisco; James Barkovich, MD, Principal Investigator — University of California, San Francisco; Pratik Mukherjee, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San francisco, San Francisco, California, United States

REFERENCES:
- [Background] Glass HC, Shaw GM, Ma C, Sherr EH. Agenesis of the corpus callosum in California 1983-2003: a population-based study. Am J Med Genet A. 2008 Oct 1;146A(19):2495-500. doi: 10.1002/ajmg.a.32418. PMID 18642362
- [Background] Tang PH, Bartha AI, Norton ME, Barkovich AJ, Sherr EH, Glenn OA. Agenesis of the corpus callosum: an MR imaging analysis of associated abnormalities in the fetus. AJNR Am J Neuroradiol. 2009 Feb;30(2):257-63. doi: 10.3174/ajnr.A1331. Epub 2008 Nov 6. PMID 18988682
- [Background] Travaglini L, Brancati F, Attie-Bitach T, Audollent S, Bertini E, Kaplan J, Perrault I, Iannicelli M, Mancuso B, Rigoli L, Rozet JM, Swistun D, Tolentino J, Dallapiccola B, Gleeson JG, Valente EM; International JSRD Study Group; Zankl A, Leventer R, Grattan-Smith P, Janecke A, D'Hooghe M, Sznajer Y, Van Coster R, Demerleir L, Dias K, Moco C, Moreira A, Kim CA, Maegawa G, Petkovic D, Abdel-Salam GM, Abdel-Aleem A, Zaki MS, Marti I, Quijano-Roy S, Sigaudy S, de Lonlay P, Romano S, Touraine R, Koenig M, Lagier-Tourenne C, Messer J, Collignon P, Wolf N, Philippi H, Kitsiou Tzeli S, Halldorsson S, Johannsdottir J, Ludvigsson P, Phadke SR, Udani V, Stuart B, Magee A, Lev D, Michelson M, Ben-Zeev B, Fischetto R, Benedicenti F, Stanzial F, Borgatti R, Accorsi P, Battaglia S, Fazzi E, Giordano L, Pinelli L, Boccone L, Bigoni S, Ferlini A, Donati MA, Caridi G, Divizia MT, Faravelli F, Ghiggeri G, Pessagno A, Briguglio M, Briuglia S, Salpietro CD, Tortorella G, Adami A, Castorina P, Lalatta F, Marra G, Riva D, Scelsa B, Spaccini L, Uziel G, Del Giudice E, Laverda AM, Ludwig K, Permunian A, Suppiej A, Signorini S, Uggetti C, Battini R, Di Giacomo M, Cilio MR, Di Sabato ML, Leuzzi V, Parisi P, Pollazzon M, Silengo M, De Vescovi R, Greco D, Romano C, Cazzagon M, Simonati A, Al-Tawari AA, Bastaki L, Megarbane A, Sabolic Avramovska V, de Jong MM, Stromme P, Koul R, Rajab A, Azam M, Barbot C, Martorell Sampol L, Rodriguez B, Pascual-Castroviejo I, Teber S, Anlar B, Comu S, Karaca E, Kayserili H, Yuksel A, Akcakus M, Al Gazali L, Sztriha L, Nicholl D, Woods CG, Bennett C, Hurst J, Sheridan E, Barnicoat A, Hennekam R, Lees M, Blair E, Bernes S, Sanchez H, Clark AE, DeMarco E, Donahue C, Sherr E, Hahn J, Sanger TD, Gallager TE, Dobyns WB, Daugherty C, Krishnamoorthy KS, Sarco D, Walsh CA, McKanna T, Milisa J, Chung WK, De Vivo DC, Raynes H, Schubert R, Seward A, Brooks DG, Goldstein A, Caldwell J, Finsecke E, Maria BL, Holden K, Cruse RP, Swoboda KJ, Viskochil D. Expanding CEP290 mutational spectrum in ciliopathies. Am J Med Genet A. 2009 Oct;149A(10):2173-80. doi: 10.1002/ajmg.a.33025. PMID 19764032
- [Background] Edwards TJ, Sherr EH, Barkovich AJ, Richards LJ. Clinical, genetic and imaging findings identify new causes for corpus callosum development syndromes. Brain. 2014 Jun;137(Pt 6):1579-613. doi: 10.1093/brain/awt358. Epub 2014 Jan 28. PMID 24477430
- [Background] Johnson-Kerner B, Snijders Blok L, Suit L, Thomas J, Kleefstra T, Sherr EH. DDX3X-Related Neurodevelopmental Disorder. 2020 Aug 27. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK561282/ PMID 32852922
- [Background] Owen JP, Li YO, Ziv E, Strominger Z, Gold J, Bukhpun P, Wakahiro M, Friedman EJ, Sherr EH, Mukherjee P. The structural connectome of the human brain in agenesis of the corpus callosum. Neuroimage. 2013 Apr 15;70:340-55. doi: 10.1016/j.neuroimage.2012.12.031. Epub 2012 Dec 23. PMID 23268782
- [Background] Lau YC, Hinkley LB, Bukshpun P, Strominger ZA, Wakahiro ML, Baron-Cohen S, Allison C, Auyeung B, Jeremy RJ, Nagarajan SS, Sherr EH, Marco EJ. Autism traits in individuals with agenesis of the corpus callosum. J Autism Dev Disord. 2013 May;43(5):1106-18. doi: 10.1007/s10803-012-1653-2. PMID 23054201
- [Background] Bina R, Matalon D, Fregeau B, Tarsitano JJ, Aukrust I, Houge G, Bend R, Warren H, Stevenson RE, Stuurman KE, Barkovich AJ, Sherr EH. De novo variants in SUPT16H cause neurodevelopmental disorders associated with corpus callosum abnormalities. J Med Genet. 2020 Jul;57(7):461-465. doi: 10.1136/jmedgenet-2019-106193. Epub 2020 Jan 10. PMID 31924697
- [Background] Fregeau B, Kim BJ, Hernandez-Garcia A, Jordan VK, Cho MT, Schnur RE, Monaghan KG, Juusola J, Rosenfeld JA, Bhoj E, Zackai EH, Sacharow S, Baranano K, Bosch DGM, de Vries BBA, Lindstrom K, Schroeder A, James P, Kulch P, Lalani SR, van Haelst MM, van Gassen KLI, van Binsbergen E, Barkovich AJ, Scott DA, Sherr EH. De Novo Mutations of RERE Cause a Genetic Syndrome with Features that Overlap Those Associated with Proximal 1p36 Deletions. Am J Hum Genet. 2016 May 5;98(5):963-970. doi: 10.1016/j.ajhg.2016.03.002. Epub 2016 Apr 14. PMID 27087320
- [Result] Sherr EH, Owen R, Albertson DG, Pinkel D, Cotter PD, Slavotinek AM, Hetts SW, Jeremy RJ, Schilmoeller G, Schilmoeller K, Wakahiro M, Barkovich AJ. Genomic microarray analysis identifies candidate loci in patients with corpus callosum anomalies. Neurology. 2005 Nov 8;65(9):1496-8. doi: 10.1212/01.wnl.0000183066.09239.b6. PMID 16275846
- [Result] Hetts SW, Sherr EH, Chao S, Gobuty S, Barkovich AJ. Anomalies of the corpus callosum: an MR analysis of the phenotypic spectrum of associated malformations. AJR Am J Roentgenol. 2006 Nov;187(5):1343-8. doi: 10.2214/AJR.05.0146. PMID 17056927
- [Result] Paul LK, Brown WS, Adolphs R, Tyszka JM, Richards LJ, Mukherjee P, Sherr EH. Agenesis of the corpus callosum: genetic, developmental and functional aspects of connectivity. Nat Rev Neurosci. 2007 Apr;8(4):287-99. doi: 10.1038/nrn2107. PMID 17375041
- [Result] Li J, Shivakumar S, Wakahiro M, Mukherjee P, Barkovich AJ, Slavotinek A, Sherr EH. Agenesis of the corpus callosum, optic coloboma, intractable seizures, craniofacial and skeletal dysmorphisms: an autosomal recessive disorder similar to Temtamy syndrome. Am J Med Genet A. 2007 Aug 15;143A(16):1900-5. doi: 10.1002/ajmg.a.31855. PMID 17632789
- [Result] Boland E, Clayton-Smith J, Woo VG, McKee S, Manson FD, Medne L, Zackai E, Swanson EA, Fitzpatrick D, Millen KJ, Sherr EH, Dobyns WB, Black GC. Mapping of deletion and translocation breakpoints in 1q44 implicates the serine/threonine kinase AKT3 in postnatal microcephaly and agenesis of the corpus callosum. Am J Hum Genet. 2007 Aug;81(2):292-303. doi: 10.1086/519999. Epub 2007 Jun 13. PMID 17668379
- [Result] Wahl M, Strominger Z, Jeremy RJ, Barkovich AJ, Wakahiro M, Sherr EH, Mukherjee P. Variability of homotopic and heterotopic callosal connectivity in partial agenesis of the corpus callosum: a 3T diffusion tensor imaging and Q-ball tractography study. AJNR Am J Neuroradiol. 2009 Feb;30(2):282-9. doi: 10.3174/ajnr.A1361. Epub 2008 Nov 11. PMID 19001538
- [Result] Nakata Y, Barkovich AJ, Wahl M, Strominger Z, Jeremy RJ, Wakahiro M, Mukherjee P, Sherr EH. Diffusion abnormalities and reduced volume of the ventral cingulum bundle in agenesis of the corpus callosum: a 3T imaging study. AJNR Am J Neuroradiol. 2009 Jun;30(6):1142-8. doi: 10.3174/ajnr.A1527. Epub 2009 Feb 26. PMID 19246528
- [Result] Wahl M, Li YO, Ng J, Lahue SC, Cooper SR, Sherr EH, Mukherjee P. Microstructural correlations of white matter tracts in the human brain. Neuroimage. 2010 Jun;51(2):531-41. doi: 10.1016/j.neuroimage.2010.02.072. Epub 2010 Mar 4. PMID 20206699
- [Result] Wahl M, Strominger ZA, Wakahiro M, Jeremy RJ, Mukherjee P, Sherr EH. Diffusion tensor imaging of Aicardi syndrome. Pediatr Neurol. 2010 Aug;43(2):87-91. doi: 10.1016/j.pediatrneurol.2010.03.005. PMID 20610117
- [Result] O'Driscoll MC, Black GC, Clayton-Smith J, Sherr EH, Dobyns WB. Identification of genomic loci contributing to agenesis of the corpus callosum. Am J Med Genet A. 2010 Sep;152A(9):2145-59. doi: 10.1002/ajmg.a.33558. PMID 20683985
- See also: Click here for more information about this study: Agenesis of the Corpus Callosum, Genetics and Clinical features — http://brain.ucsf.edu/research-studies
- See also: National Organization of the Disorders of the Corpus Callosum (a non-profit corporation) — http://www.nodcc.org/
- See also: UCSF Clinical Trials — https://clinicaltrials.ucsf.edu/trial/NCT00305305